CLINICAL TRIAL: NCT00086996
Title: Oxaliplatin (NSC-266046) Plus Protracted Infusion 5-Fluorouracil And Radiation For Potentially Curable Esophageal Cancer: A Phase II Trial With Molecular Correlates
Brief Title: S0356 Oxaliplatin, 5-FU, Radiation Therapy (RT), Surgery for Pts With Stage II or III Cancer of Esophagus or Gastroesophageal (GE) Junction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000371963; U10CA032102 (NIH); S0356 (Other: SWOG)
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Results first posted 2012-04-03 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2013-09

CONDITIONS: Esophageal Cancer
Keywords: adenocarcinoma of the esophagus; stage II esophageal cancer; stage III esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus | interventions — Fluorouracil; Oxaliplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemo Plus RT, Surgery, Chemo (Experimental): neoadjuvant fluorouracil, oxaliplatin and radiation therapy followed by conventional surgery and adjuvant fluoruracil and oxaliplatin
  Interventions: Drug: fluorouracil; Drug: oxaliplatin; Procedure: conventional surgery; Radiation: radiation therapy

INTERVENTIONS:
Drug: fluorouracil — Before surgery: 180 mg/m2/day by 24-hour infusion days 8 through 43. After surgery:180 mg/m2/day by 24-hour infusion days 1 through 36.
  Other Names: 5-FU
Drug: oxaliplatin — Before surgery: 85 mg/m2 by 2-hour IV infusion days 1, 15, and 29. After surgery: 85 mg/m2 by 2-hour IV infusion days 1, 15, and 29.
  Other Names: eloxatin
Procedure: conventional surgery — The surgical technique will depend upon the location and extent of tumor and individual surgeon preference.
Radiation: radiation therapy — Starting Day 8, patients will be treated 5 days/week at 180 centigray (cGy)/day times 25 fractions to a total dose of 4,500 cGy.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as oxaliplatin and fluorouracil, work in different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Oxaliplatin and fluorouracil may make tumor cells more sensitive to radiation therapy and may kill more tumor cells. Giving chemotherapy and radiation therapy before surgery may shrink the tumor so that it can be removed.

PURPOSE: This phase II trial is studying how well giving oxaliplatin together with fluorouracil and radiation therapy works in treating patients who are undergoing surgery for stage II or stage III cancer of the esophagus or gastroesophageal junction.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the pathologic complete response probability in patients with stage II or III adenocarcinoma of the esophagus or gastroesophageal junction treated with neoadjuvant oxaliplatin, fluorouracil, and radiotherapy followed by definitive surgical resection.

Secondary

* Determine the frequency and severity of toxic effects associated with this neoadjuvant regimen in these patients.
* Determine the overall survival and progression-free survival of patients treated with this regimen.

Exploratory Analyses (subject to funding availability)

* Correlate, preliminarily, initial messenger ribonucleic acid (mRNA) levels of the genes for thymidylate synthase (TS), γ-glutamyl transpeptidase (γGT), γ-glutamyl cysteine (γ-GCS), DNA excision repair cross-complementing (ERCC-1), and xeroderma pigmentosum (XPA) with response and survival of patients treated with this regimen.
* Correlate, preliminarily, the mRNA levels of TS, γGT, γ-GCS, ERCC-1, and XPA before and after treatment with this regimen with survival of these patients.
* Correlate, preliminarily, specific genetic polymorphisms of TS and ERCC-1 with tumor response and overall survival of patients treated with this regimen.

OUTLINE: This is a multicenter study.

* Neoadjuvant chemoradiotherapy: Patients receive oxaliplatin IV over 2 hours on days 1, 15, and 29 and fluorouracil (5-FU) IV continuously on days 8-43. Beginning on day 8, patients also undergo radiotherapy once daily, 5 days a week, for 5 weeks.
* Surgery: Patients with stable disease or better undergo surgical resection 4-10 weeks after completion of chemoradiotherapy.
* Adjuvant chemotherapy: Beginning 4-10 weeks after surgery, patients receive chemotherapy comprising oxaliplatin IV over 2 hours on days 1, 15, and 29 and 5-FU IV continuously on days 1-36.

Treatment continues in the absence of unacceptable toxicity or disease progression.

Patients are followed every 3 months for 1 year and then every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 45-85 patients will be accrued for this study within 17-21 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary adenocarcinoma of the thoracic esophagus or gastroesophageal junction

  * No recurrent disease
  * Primary esophageal tumor at least 20 cm below the incisors (if < 26 cm below the incisors, a bronchoscopy must be performed and cytology must be negative)
  * Esophageal disease confined to esophagus and peri-esophageal soft tissue
  * Gastroesophageal junction disease extending ≤ 2 cm into the gastric cardia
* Clinical stage II or III disease by CT scan or MRI

  * If no esophageal mass is detected by these methods, esophageal endoscopic ultrasound is required to determine stage
  * Positron-emission tomography scan is required to confirm stage
* Measurable or non-measurable disease by x-ray, scanning, or physical examination
* No celiac axis nodes ≥ 1.5 cm

  * Measurable regional lymph nodes ≥ 1.5 cm at stations 2-10=N1 OR subdiaphragmatic lymph nodes at stations 15-19 ≤ 1.5 cm by CT scan or MRI allowed
  * Palpable supraclavicular lymph nodes must be free of metastatic esophageal cancer by biopsy

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* White blood cell (WBC) count ≥ 3,000/mm^3
* Hemoglobin ≥ 10.0 g/dL (transfusion allowed)

Hepatic

* Albumin ≥ 3 g/dL
* Bilirubin normal

Renal

* Creatinine ≤ 1.5 times upper limit of normal

Cardiovascular

* No myocardial infarction or cerebrovascular event within the past 6 months

Pulmonary

* No active pneumonia or inflammatory lung infiltrate

Other

* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No peripheral neuropathy ≥ grade 2
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for esophageal cancer

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy for esophageal cancer
* No concurrent intensity-modulated radiotherapy

Surgery

* No prior surgical resection or attempted surgical resection of esophageal cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2004-09; Primary Completion 2009-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence P. Leichman, MD, Study Chair — Desert Regional Medical Center Comprehensive Cancer Center; Charles R. Thomas, MD, Study Chair — OHSU Knight Cancer Institute
Locations (143):
- United States (143):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Providence Cancer Center, Anchorage, Alaska
  - Highlands Oncology Group - Springdale, Bentonville, Arkansas
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Medical Center, Castro Valley, California
  - Valley Medical Oncology Consultants - Castro Valley, Castro Valley, California
  - Valley Medical Oncology, Fremont, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Breast Surgeons, Incorporated, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Larry G Strieff MD Medical Corporation, Oakland, California
  - Tom K Lee, Incorporated, Oakland, California
  - Desert Regional Medical Center Comprehensive Cancer Center, Palm Springs, California
  - Valley Care Medical Center, Pleasanton, California
  - Valley Medical Oncology Consultants - Pleasanton, Pleasanton, California
  - University of California Davis Cancer Center, Sacramento, California
  - Doctors Medical Center - San Pablo Campus, San Pablo, California
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Olathe Cancer Center, Olathe, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - St. Francis Comprehensive Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Metro Health Hospital, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Missouri Regional Cancer Center at Southeast Missouri Hospital, Gape Girardeau, Missouri
  - St. John's Regional Medical Center, Joplin, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Frontier Cancer Center, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Tucker Center for Cancer Care at Orange Regional Medical Center, Middletown, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Moses Cone Regional Cancer Center at Wesley Long Community Hospital, Greensboro, North Carolina
  - Annie Penn Cancer Center, Reidsville, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - AnMed Cancer Center, Anderson, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Christine LaGuardia Phillips Cancer Center at Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - CCOP - Scott and White Hospital, Temple, Texas
  - American Fork Hospital, American Fork, Utah
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Southwest Virginia Regional Cancer Center at Wellmonth Health, Norton, Virginia
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Rockwood Clinic Cancer Treatment Center, Spokane, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Result] Leichman L, Goldman BH, Benedetti JK, et al.: Oxaliplatin (OXP) plus protracted infusion 5-fluorouracil (PIFU) and external beam radiation (EBRT) prior to surgery (S) for potentially curable esophageal adenocarcinoma (EA): A Southwest Oncology Group (SWOG) phase II trial with molecular correlates (S0356). [Abstract] J Clin Oncol 27 (Suppl 15): A-4513, 2009.
- [Derived] Leichman LP, Goldman BH, Bohanes PO, Lenz HJ, Thomas CR, Billingsley KG, Corless CL, Iqbal S, Gold PJ, Benedetti JK, Danenberg KD, Blanke CD. S0356: a phase II clinical and prospective molecular trial with oxaliplatin, fluorouracil, and external-beam radiation therapy before surgery for patients with esophageal adenocarcinoma. J Clin Oncol. 2011 Dec 1;29(34):4555-60. doi: 10.1200/JCO.2011.36.7490. Epub 2011 Oct 24. PMID 22025151

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemo Plus RT, Surgery, Chemo: * Neoadjuvant chemoradiotherapy: Patients receive oxaliplatin 85 mg/m^2 by 2-hour IV infusion days 1, 15, and 29 and fluorouracil (5-FU) 180 mg/m^2/day infusion continuously on days 8-43. Beginning on day 8, patients also undergo radiotherapy at 180 centigray (cGy)/day, 5 days a week, for 5 weeks to a total dose of 4,500 cGy.
  * Surgery: Patients with stable disease or better undergo surgical resection 4-10 weeks after completion of chemoradiotherapy. The surgical technique will depend upon the location and extent of tumor and individual surgeon preference.
  * Adjuvant chemotherapy: Beginning 4-10 weeks after surgery, patients receive chemotherapy comprising oxaliplatin 85 mg/m^2 by 2-hour IV infusion days 1, 15, and 29 and 5-FU 180 mg/m^2/day by 24-hour infusion continuously on days 1-36.
Period: Overall Study
Arm/Group | Chemo Plus RT, Surgery, Chemo
Started | 98
Eligible | 93
Eligible and Began Protocol Therapy | 93
Completed | 34
Not Completed | 64
Not completed — Adverse Event | 29
Not completed — Death | 4
Not completed — progression/relapse | 7
Not completed — Withdrawal by Subject | 13
Not completed — Other | 6
Not completed — not eligible | 5

BASELINE CHARACTERISTICS:
Arm/Group | Chemo Plus RT, Surgery, Chemo
Number analyzed (Participants) | 93
Age Continuous [Median (Full Range); unit: participants] — Of eligible patients
  participants | 62.2 [41.6 to 83.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 87
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 86
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 86
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Pathological Complete Response
Description: Complete pathologic response assessed after chemoradiotherapy and surgery, defined as no evidence of residual disease on path review. Patients who did not receive surgery are assumed to have not responded.
Time Frame: 10-16 weeks after beginning study treatment
Population: Eligible patients
Measure: Number; unit: participants
Arm/Group | Chemo Plus RT, Surgery, Chemo
Number analyzed (Participants) | 93
participants | 26

2. Secondary Outcome: Number of Patients With Grade 3 Through 5 Adverse Events That Are Related to Study Drug
Description: Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Up to 3 years
Population: Eligible patients who received any treatment and were assessed for toxicity were included in the adverse event summaries. Any Common Terminology Criteria for Adverse Events (CTCAE) v3.0 event of Grade 3 (severe), Grade 4 (life threatening), or Grade 5 (fatal) which were deemed to be related to protocol treatment are included.
Measure: Number; unit: Participants
Arm/Group | Chemo Plus RT, Surgery, Chemo
Number analyzed (Participants) | 93
Participants
  Adult respiratory distress syndrome (ARDS) | 4
  Anorexia | 15
  CNS cerebrovascular ischemia | 1
  Calcium, serum-low (hypocalcemia) | 2
  Cardiac troponin T (cTnT) | 1
  Cardiac-ischemia/infarction | 1
  Chyle or lymph leakage | 1
  Confusion | 1
  Cough | 1
  Creatinine | 1
  Dehydration | 3
  Diarrhea | 12
  Distention/bloating, abdominal | 1
  Dysphagia (difficulty swallowing) | 4
  Dyspnea (shortness of breath) | 3
  Esophagitis | 3
  Fatigue (asthenia, lethargy, malaise) | 14
  Febrile neutropenia | 1
  Fever in absence of neutropenia, ANC lt1.0x10e9/L | 1
  Fistula, GI - Oral cavity | 1
  Gastrointestinal-Other (Specify) | 1
  Glucose, serum-high (hyperglycemia) | 3
  Heartburn/dyspepsia | 1
  Hemoglobin | 4
  Hypotension | 1
  Hypoxia | 6
  Inf (clin/microbio) w/Gr 3-4 neuts - Lung | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - Blood | 2
  Inf w/normal ANC or Gr 1-2 neutrophils - Lung | 3
  Inf w/normal ANC or Gr 1-2 neutrophils - Perit cav | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - Wound | 4
  Infection with unknown ANC - Blood | 1
  Infection with unknown ANC - Lung (pneumonia) | 2
  Infection with unknown ANC - Wound | 1
  Leak (including anastomotic), GI - Esophagus | 1
  Leukocytes (total WBC) | 2
  Lymphopenia | 10
  Mood alteration - anxiety | 1
  Mucositis/stomatitis (clinical exam) - Esophagus | 1
  Mucositis/stomatitis (clinical exam) - Oral cavity | 4
  Mucositis/stomatitis (functional/symp) - Esophagus | 5
  Mucositis/stomatitis (functional/symp) - Oral cav | 2
  Muscle weakness, not d/t neuropathy - body/general | 1
  Nausea | 11
  Necrosis, GI - Stomach | 1
  Neutrophils/granulocytes (ANC/AGC) | 1
  Obstruction, GI - Esophagus | 1
  Pain - Abdomen NOS | 1
  Pain - Pain NOS | 1
  Pericardial effusion (non-malignant) | 4
  Platelets | 2
  Pleural effusion (non-malignant) | 3
  Pneumonitis/pulmonary infiltrates | 3
  Potassium, serum-low (hypokalemia) | 4
  Pulmonary/Upper Respiratory-Other (Specify) | 3
  Renal failure | 1
  SVT and nodal arrhythmia - Atrial fibrillation | 2
  SVT and nodal arrhythmia - Sinus tachycardia | 1
  Skin breakdown/decubitus ulcer | 1
  Sodium, serum-low (hyponatremia) | 5
  Stricture/stenosis (incl anastomotic), Esophagus | 2
  Syncope (fainting) | 1
  Thrombosis/thrombus/embolism | 2
  Typhlitis (cecal inflammation) | 1
  Vomiting | 7
  Weight loss | 13
  Wound complication, non-infectious | 1

3. Secondary Outcome: Overall Survival
Description: Measured from time of registration to death, or last contact date
Time Frame: 0-5 years
Population: eligible patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemo Plus RT, Surgery, Chemo
Number analyzed (Participants) | 93
months | 28.3 [22.4 to 52.4]

4. Secondary Outcome: Progression-free Survival
Description: measured from date of registration to time of first documentation of progression by Response Evaluation Criteria in Solid Tumors (RECIST), death, or last contact date.
Time Frame: 0-3 years
Population: eligible patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemo Plus RT, Surgery, Chemo
Number analyzed (Participants) | 93
months | 19.7 [14.7 to 28.3]

ADVERSE EVENTS:
Time Frame: Up to 3 years
Arm/Group | Chemo Plus RT, Surgery, Chemo
Serious Adverse Events (participants affected / at risk) | 7/93
Other Adverse Events (participants affected / at risk) | 93/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemo Plus RT, Surgery, Chemo (N=93)
Cardiac-ischemia/infarction (Cardiac disorders) | 1
Pericardial effusion (non-malignant) (Cardiac disorders) | 1
SVT and nodal arrhythmia - Atrial fibrillation (Cardiac disorders) | 1
Typhlitis (cecal inflammation) (Gastrointestinal disorders) | 1
Inf (clin/microbio) w/Gr 3-4 neuts - Lung (Infections and infestations) | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Blood (Infections and infestations) | 1
Cardiac troponin I (cTnI) (Investigations) | 1
Adult respiratory distress syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Thrombosis/thrombus/embolism (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chemo Plus RT, Surgery, Chemo (N=93)
Hemoglobin (Blood and lymphatic system disorders) | 67
SVT and nodal arrhythmia - Atrial fibrillation (Cardiac disorders) | 16
SVT and nodal arrhythmia - Sinus tachycardia (Cardiac disorders) | 8
Constipation (Gastrointestinal disorders) | 28
Diarrhea (Gastrointestinal disorders) | 59
Distention/bloating, abdominal (Gastrointestinal disorders) | 5
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 40
Esophagitis (Gastrointestinal disorders) | 10
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 5
Gastrointestinal-Other (Specify) (Gastrointestinal disorders) | 8
Heartburn/dyspepsia (Gastrointestinal disorders) | 18
Mucositis/stomatitis (clinical exam) - Esophagus (Gastrointestinal disorders) | 5
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 18
Mucositis/stomatitis (functional/symp) - Esophagus (Gastrointestinal disorders) | 16
Mucositis/stomatitis (functional/symp) - Oral cav (Gastrointestinal disorders) | 13
Nausea (Gastrointestinal disorders) | 76
Pain - Abdomen NOS (Gastrointestinal disorders) | 13
Pain - Esophagus (Gastrointestinal disorders) | 17
Stricture/stenosis (incl anastomotic), Esophagus (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 42
Fatigue (asthenia, lethargy, malaise) (General disorders) | 77
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 19
Pain - Chest/thorax NOS (General disorders) | 9
Pain-Other (Specify) (General disorders) | 7
Inf w/normal ANC or Gr 1-2 neutrophils - Lung (Infections and infestations) | 5
Inf w/normal ANC or Gr 1-2 neutrophils - Wound (Infections and infestations) | 8
Leak (including anastomotic), GI - Esophagus (Injury, poisoning and procedural complications) | 5
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 17
AST, SGOT (Investigations) | 16
Alkaline phosphatase (Investigations) | 23
Bilirubin (hyperbilirubinemia) (Investigations) | 11
Creatinine (Investigations) | 11
Leukocytes (total WBC) (Investigations) | 37
Lymphopenia (Investigations) | 15
Metabolic/Laboratory-Other (Specify) (Investigations) | 6
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 12
Platelets (Investigations) | 43
Weight loss (Investigations) | 53
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 31
Anorexia (Metabolism and nutrition disorders) | 56
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 29
Dehydration (Metabolism and nutrition disorders) | 25
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 36
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 6
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 5
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 23
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 29
Pain - Back (Musculoskeletal and connective tissue disorders) | 5
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 6
Dizziness (Nervous system disorders) | 13
Neuropathy: sensory (Nervous system disorders) | 55
Pain - Head/headache (Nervous system disorders) | 5
Taste alteration (dysgeusia) (Nervous system disorders) | 14
Insomnia (Psychiatric disorders) | 10
Mood alteration - anxiety (Psychiatric disorders) | 11
Mood alteration - depression (Psychiatric disorders) | 13
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 5
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 19
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 13
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 11
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 13
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 8
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 8
Pulmonary/Upper Respiratory-Other (Specify) (Respiratory, thoracic and mediastinal disorders) | 5
Rash/desquamation (Skin and subcutaneous tissue disorders) | 9
Hypotension (Vascular disorders) | 9
Thrombosis/thrombus/embolism (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No